CLINICAL TRIAL: NCT06293027
Title: Establishing Novel Functional Biomarkers for Fragile X Syndrome
Brief Title: Optical Imaging as a Tool for Monitoring Brain Function in Fragile X Syndrome
Status: Recruiting | Type: Observational
Sponsor: IRCCS Fondazione Stella Maris (Other)
Responsible Party: Sponsor
Other Study IDs: IMAGINER FXS
Record Dates: First submitted 2024-02-20; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Fragile X Syndrome
MeSH Terms: conditions — Fragile X Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FXS affected individuals: Individuals with genetic diagnosis of FXS.
- Neurotypical controls: Healthy volunteers without known health or medical issues.

SUMMARY:
The objective of this project is to explore the potential of functional near- infrared spectroscopy (fNIRS) as innovative functional biomarker for clinical trial readiness in Fragile X Syndrome (FXS) that is still without cure. The limited availability of objective and quantitative biomarkers to monitor brain function poses challenges to advancing therapeutic research. With clinical trials on the horizon, the need for precise measurement to evaluate treatment efficacy is pressing. The investigators seek to address this gap by assessing the prognostic reliability of both resting and task- evoked fNIRS. The primary objectives of this pilot study are: 1. to determine the feasibility of fNIRS in individuals with FXS; 2. to collect pilot data on individuals with FXS to determine the patterns of cerebral oxygen consumption as measured by fNIRS; 3. to compare cerebral oxygen consumption changes at rest and from visual/auditory tasks in affected individuals versus age-appropriate healthy volunteers. The secondary objectives of this study are: 1. to correlate cerebral oxygen consumption changes from visual/auditory task in affected individuals to other measures of disease state (e.g., neuropsychological assessment, disease- specific severity rating scales); 2. to examine test-retest reliability of our fNIRS measures in both affected individuals and healthy controls.

DETAILED DESCRIPTION:
This is a non-profit study of a cohort of patients with genetically determined Fragile X Syndrome and age-matched healthy controls. The design of the study is observational, case-control. An imaging session using fNIRS (NIRSport2, NIRx Technologies) will be conducted during the visits scheduled for the individual participants. Participants will be assessed for optimal placement of the fNIRS probe on the head through measurement of the fiducial points on the scalp. With the NIRx NIRSPort2 system, the near- infrared sources and detectors are situated in a fabric cap resembling a swim cap that is applied like a hat and secured in place by a velcro chin strap.

Once the probe is placed, fNIRS will be measured during a passive viewing/ listening task administered on a computer. The montage consists of 8 red light-sources operating at 760 nm and 850 nm, and 7 detectors which can be easily placed into a textile EEG cap (EASYCAP, Herrsching, Germany, size according to head circumference). The systems that are utilized have been selected to be very child-friendly systems, involving no cleaning or abrasion of the scalp preparation and rapid application. Application procedures have been designed to minimize any discomfort to the participant. In total, these measurements should take 30-40 minutes to complete (including application of the NIRS cap). Alongside fNIRS, neuropsychological assessments of affected individuals patients will be conducted. The following outcome measures will be collected assessing: i) cognitive performance (Leiter International Performance Scale, 3rd edition, PPVT-5, simple reasoning tasks on tablets and Vineland Adaptive Behaviour Scale); ii) behavioural disorder (BASC-3, ABC-2 scales and BRIEF); iii) autistic-like features (SRS-2 and PPD- MRS). The cognitive tasks were chosen to be adapted to the cognitive deficit of affected individuals. A task on tablets with minimal verbal instruction will allow to assess reasoning abilities in severe to moderate ID patients that could not perform classical Wechsler scale (IQ test). Healthy controls will be asked to return 8-12 weeks post their initial visit to undergo repeat fNIRS testing for the purposes of examining test-retest reliability of the fNIRS measurement. If their schedule allows, affected individuals will also undergo repeat fNIRS testing. fNIRS is safe, non-invasive and generally well tolerated. The information obtained from this study will help identify outcome measures for drug testing in future therapeutic trials.

ELIGIBILITY:
Inclusion Criteria:

FXS participants:

* Age criteria: Between ages 2 years to 50 years old, inclusive at time of enrollment
* Diagnosed with FXS with a previously identified pathogenic or likely pathogenic variant in the FMR1 gene.
* Must also meet the diagnostic criteria for FXS.
* Male

Typically developing participants:

* Age criteria: Between ages 2 years to 50 years old, inclusive at time of enrollment
* Age- and sex-matched to the FXS participants
* No underlying genetic diagnosis or past/chronic medical condition associated with increased risk for autism spectrum disorder (ASD) and/or ID
* Typical neurodevelopment for age (no established diagnosis or clinical suspicion for ASD or ID)

Exclusion Criteria:

For FXS and Typically developing participants:

* Unwilling or unable to comply with study procedures and assessments
* Contraindications to fNIRS, such as uncooperative or destructive behaviors preventing lead placement or capture by fNIRS equipment
* Traumatic loss of consciousness in the last year
* Has taken an investigational drug as part of another research study, within 30 days prior to study enrollment
* If participant is judged by the PI or Sub-I to be inappropriate for the study for any reason

For Typically developing participants:

* Known or suspected cognitive impairment
* Known history of MRI abnormality
* Current use of psychotropic medications

Min Age: 2 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Fragile X syndrome (FXS) is the most commonly inherited form of mental retardation and developmental disabilities, affecting 1 in 4000 individuals. The phenotype of FXS involves mental retardation or learning disabilities, social deficit, anxiety, attention deficit, impulsivity, hyperarousal, mood instability, inflexibility, prominent ears, long face, and hyperextensible finger joints. There is no effective treatment for FXS, and the standard of care include therapies that help minimise the symptoms of the condition.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Resting-state functional connectivity | 3 years
  The comparison of resting-state fNIRS signal between affected individuals and healthy controls will allow to detect potential alterations of spontaneous brain activity and functional connectivity
Amplitude of sensory-evoked hemodynamic responses | 3 years
  The analysis of the amplitude of sensory-evoked fNIRS signal will allow to assess whether this parameter is able to discriminate between affected individuals and healthy controls. The signal latency will be analysed as well.

SECONDARY OUTCOMES:
Correlation between neurophysiology endpoints and the response on neuropsychological scale. | 3 years
  The correlation analysis will allow to understand whether alterations of functional connectivity and/or sensory-evoked responses can be predictive of the severity of symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Stella Maris, Tirrenia, Tuscany, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mazziotti R, Scaffei E, Conti E, Marchi V, Rizzi R, Cioni G, Battini R, Baroncelli L. The amplitude of fNIRS hemodynamic response in the visual cortex unmasks autistic traits in typically developing children. Transl Psychiatry. 2022 Feb 8;12(1):53. doi: 10.1038/s41398-022-01820-5. PMID 35136021
- [Background] Scaffei E, Mazziotti R, Conti E, Costanzo V, Calderoni S, Stoccoro A, Carmassi C, Tancredi R, Baroncelli L, Battini R. A Potential Biomarker of Brain Activity in Autism Spectrum Disorders: A Pilot fNIRS Study in Female Preschoolers. Brain Sci. 2023 Jun 14;13(6):951. doi: 10.3390/brainsci13060951. PMID 37371429